CLINICAL TRIAL: NCT05699798
Title: Comparison of the Efficacy of Instrument-assisted Soft Tissue Mobilization and Extracorporeal Shock Wave Therapy in Myofascial Pain Syndrome
Brief Title: The Aim of This Study is to Compare the Effects of Instrument-assisted Soft Tissue Mobilization (IASTM) and Extracorporeal Shock Wave Therapy (ESWT) Used in Myofascial Pain Syndrome (MPS) and to Determine Whether They Are Superior to Conservative Treatment (CT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, şeyda candeniz, Instructor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: candeniz-001
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Myofascial Pain Syndrome
Keywords: IASTM; ESWT; Myofascial Pain Syndrome; Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Conservative Treatment; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conservative Treatment (CT) (Experimental): Includes Hotpack, TENS, Ultrasound and home exercise programs. HP, US and TENS applications were applied for 3 weeks, with a total of 15 sessions, 5 sessions per week. HP application for 20 minutes, ultrasound for 5 minutes and TENS for 20 minutes were applied to the patients. The CT protocol was applied to all three groups in the same way.
  Interventions: Other: Conservative Treatment (CT)
- Instrument Assisted Soft Tissue Mobilization (IASTM) (Experimental): Includes Hotpack, TENS, Ultrasound, home exercise programs and Instrument-assisted Soft Tissue Mobilization Technique. The IASTM therapy was applied for three weeks, two sessions per week, for a total of 6 sessions.
  Interventions: Other: Instrument-assisted Soft Tissue Mobilization (IASTM)
- Extracorporeal Shock Wave Therapy (ESWT) (Experimental): Includes Hotpack, TENS, Ultrasound, home exercise programs and Extracorporeal Shock Wave Therapy treatment. The ESWT therapy was applied for three weeks, two sessions per week, for a total of 6 sessions.
  Interventions: Other: Extracorporeal Shock Wave Therapy (ESWT)

INTERVENTIONS:
Other: Conservative Treatment (CT) — Conservative treatment (HP, US, TENS) was applied for 3 weeks, with 5 sessions per week, a total of 15 sessions.
  Arms: Conservative Treatment (CT)
Other: Instrument-assisted Soft Tissue Mobilization (IASTM) — IASTM was performed only on the neck and upper back muscles on the aching side using the sweep technique on the origo and insertion lines. A total of 6 sessions were applied, two sessions per week for 3 weeks.
  Conservative treatment (HP, US, TENS) was applied for 3 weeks, with 5 sessions per week, a total of 15 sessions.
  Arms: Instrument Assisted Soft Tissue Mobilization (IASTM)
Other: Extracorporeal Shock Wave Therapy (ESWT) — ESWT therapy was applied on the muscle with active trigger point, at 1.5-2.0 bar pressure, at 10 Hz frequency, 2000 beats in each session, twice a week, in total 6 sessions.
  Conservative treatment (HP, US, TENS) was applied for 3 weeks, with 5 sessions per week, a total of 15 sessions.
  Arms: Extracorporeal Shock Wave Therapy (ESWT)

SUMMARY:
The Aim of This Study is to Compare the Effects of Instrument-assisted Soft Tissue Mobilization (IASTM) and Extracorporeal Shock Wave Therapy (ESWT) Used in Myofascial Pain Syndrome (MPS) and to Determine Whether They Are Superior to Conservative Treatment (CT). 42 Female Patients Diagnosed With MPS Were Included in the Study. The Patients Were Randomly Divided Into Three Groups of 14 People Each. CT (Hot Pack, TENS, Ultrasound) Was Applied to the First Group. CT+IASTM Was Applied to the Second Group and CT+ESWT Was Applied to the Third Group. All Groups Received Treatment for 3 Weeks (CT: 5 Sessions Per Week, 15 Sessions in Total, ESWT and IASTM: 2 Sessions Per Week, 6 Sessions in Total). Neck Stretching Exercises Were Given to All Patients as a Home Program. Before and After the Treatment, the Pain Intensity of the Patients Was Determined by Visual Analog Scale (VAS). Pressure Pain Threshold Was Measured With an Algometer. Cervical Joint Range of Motion (CROM) Was Measured With a CROM Device. Pain, Cervical Mobility, Quality of Life, and Sleep Parameters Were Evaluated With the Neck Outcome Score Questionnaire (NOOS). Depression and Anxiety Parameters Were Evaluated With the Hospital Anxiety and Depression Scale (HADS).

DETAILED DESCRIPTION:
Ethics Approval: The study started with the approval of the Ethics Committee of Gazi University Faculty of Medicine with the 30.05.2022- 427 protocol number.

Randomization:42 female patients included in the study were randomized into 3 groups.

Interventions:The first group received a Conservative Treatment (CT) program including Hotpack (HP), Ultrasound (US) and Transcutaneous Electrical Nerve Stimulation (TENS), which is routinely given in physical therapy clinics. The second group was given Instrument-Assisted Soft Tissue Mobilization (IASTM) treatment in addition to the CT we applied in the first group. Extracorporeal Shock Wave Therapy (ESWT) was applied to the third group in addition to the CT we applied in the first group. In addition, a home exercise program consisting of neck stretching exercises was given to all participants. The effects of treatments on pain severity, pressure pain threshold, cervical joint range of motion, neck mobility, sleep, activity-pain, quality of life, anxiety and depression were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* To be diagnosed with Myofascial Pain Syndrome (MPS) according to Simons diagnostic criteria (having 5 major and at least one minor criterion)
* Detection of a trigger point in the trapezius muscle
* Not receiving any treatment for MPS in the last 1 month

Exclusion Criteria:

* Serious cervical disc disorders
* Tumor
* Fibromyalgia
* Mental or psychotic disorders
* Venous insufficiency
* Active infection
* Pregnancy
* Allergic skin diseases
* Acute rheumatic diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the anatomical muscle structure and physiology of men and women are different, we only made it in women in order to eliminate this difference.
Enrollment: 42 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline
  The Pain Intensity of the patients was determined by Visual Analog Scale (VAS).The scale is scored between 0 and 10. "0" means no pain, "10" means very severe pain.
Pain Intensity | Third week (Posttreatment)
  The Pain Intensity of the patients was determined by Visual Analog Scale (VAS).The scale is scored between 0 and 10. "0" means no pain, "10" means very severe pain.
Pressure Pain Threshold | Baseline
  Pressure Pain Threshold was measured with an algometer. The algometer evaluates the patient's pain threshold and gives a numerical data.
Pressure Pain Threshold | Third week (Posttreatment)
  Pressure Pain Threshold was measured with an algometer. The algometer evaluates the patient's pain threshold and gives a numerical data.
Cervical Joint Range of Motion | Baseline
  Cervical Joint Range of Motion (ROM) was measured with a CROM Device. The degrees of flexion, extension, right rotation, left rotation, right lateral flexion, and left lateral flexion obtained during active joint movement of the cervical region were measured.
Cervical Joint Range of Motion | Third week (Posttreatment)
  Cervical Joint Range of Motion (ROM) was measured with a CROM Device. The degrees of flexion, extension, right rotation, left rotation, right lateral flexion, and left lateral flexion obtained during active joint movement of the cervical region were measured.

SECONDARY OUTCOMES:
Disability | Baseline
  Disability, Cervical Mobility, Sleep and Quality of Life parameters were evaluated with the Neck Outcome Score Questionnaire (NOOS).
Disability | Third week (Posttreatment)
  Disability, Cervical Mobility, Sleep and Quality of Life parameters were evaluated with the Neck Outcome Score Questionnaire (NOOS).
Depression and Anxiety | Baseline
  Depression and Anxiety parameters were evaluated with the Hospital Anxiety and Depression Scale (HADS).
Depression and Anxiety | Third week (Posttreatment)
  Depression and Anxiety parameters were evaluated with the Hospital Anxiety and Depression Scale (HADS).

CONTACTS AND LOCATIONS:
Overall Officials: Seyda CANDENIZ, PhD, Principal Investigator — Ankara University; Zafer GUNENDI, Prof.Dr., Study Director — Gazi University; Seyit CITAKER, Prof.Dr., Study Director — Gazi University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No